CLINICAL TRIAL: NCT01667627
Title: A Double-blind, Placebo-controlled Study to Assess the Effect of Probiotic on Symptom Relief and Indices of Micro-inflammation and Cholinergic Status in IBS Patients With Diarrhea.
Brief Title: Probiotic in Irritable Bowel Syndrome (IBS) Patients With Diarrhea
Acronym: IBS-D
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TASMC-11-RD-0491-CTIL
Record Dates: First submitted 2012-08-15; First posted 2012-08-17 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: IBS
Keywords: IBS; Probiotic; hs-CRP; Cholinergic status; Micro-inflammation
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIO-25, Probiotic-mixture (Active Comparator): Two capsules a day.
  Interventions: Dietary Supplement: Bio-25
- Placebo (Placebo Comparator): Identical to the Bio-25 capsule: same taste, same colour, same appearance
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Bio-25 — Each capsule of the multispecies probiotic combination Bio-25 consists of 25 billion live bacteria.
  Each type of bio-25 contains billions of live lactic acid bacteria in defined ratios of lyophilized Bifidobacterium breve, Bifidobacterium longum, Bifidobacterium infantis, Lactobacillus acidophilus, Lactobacillus plantarum, Lactobacillus paracasein, Lactobacillus casei, Bifidobacterium bifidum,Lactobacillus lactis, Lactobacillus rhamnosus,and Streptococcus thermophilus.
  Other Names: Probiotic
  Arms: BIO-25, Probiotic-mixture
Other: Placebo — Identical placebo
  Arms: Placebo

SUMMARY:
We present the study design of a clinical trial designed to assess the clinical effects of the multispecies probiotic combination "BIO-25" in IBS-D patients. To this aim the primary endpoints of the study will be improvement in abdominal pain and stool consistency. The study will also be designed and powered to investigate the effect of the probiotic BIO-25 on the putative inflammation-associated parameters related to microinflammation in IBS, using postulated improvements in Hs-CRP, and calprotectin as markers of that effect. Additional aims of the study will examine the possible effect of probiotic BIO-25 on the cholinergic status.

DETAILED DESCRIPTION:
Probiotic treatment in IBS is safe and effective. Probiotics have been shown to improve the anti-inflammatory/proinflammatory ratio, and may also improve intestinal motility, and the bacterial composition of the intestines. There is a substantial body of evidence in support of the use of probiotics in IBS. Probiotics appear to be particularly effective in the reduction of abdominal bloating and discomfort. The strains of the multispecies probiotic combination (BIO-25 LR) were tested and found to be beneficial in well-designed studies of IBS patients. Patients with post-infectious IBS, as well as many patients with "classic" IBS, manifest a low-grade inflammatory state that may be associated with visceral hypersensitivity and impaired motility. Probiotics may suppress this low-grade inflammation. In a recent study we found that highly sensitive CRP (hs-CRP), a serum marker of micro-inflammation, was significantly higher in patients with diarrhea-predominant IBS than healthy controls, although within normal limits in both groups. Thus, hs-CRP may serve as a marker of this low-grade, sub-clinical inflammation. If treatment with probiotic reduces the degree of low-grade inflammation in IBS, the improvement may be reflected in reduced hs-CRP levels. This study can contribute to our understanding of the pathophysiology of IBS and provide further evidence for the effectiveness of probiotic in its treatment.

ELIGIBILITY:
Inclusion Criteria:

A diagnosis of IBS-D according to the Rome III criteria, agreement to participate and the ability to sign an informed consent. Moreover, the definition of inclusion criteria is based on the FDA Draft Guidance for Clinical Evaluation of Products (add ref here). Over the two week run-in period:

* Pain Intensity: weekly average of worst abdominal pain in past 24 hours score of ≥ 3.0 on a 0 (no pain at all) to 10 (worst possible pain) point scale
* Stool Consistency: ≥30% of days/week with at least one stool ≥6 using the Bristol Stool Score (BSS, Fig. 1) (ref).

Exclusion Criteria:

1) Hyperthyroidism, 2) celiac disease 3) pregnancy, 4) other gastrointestinal diagnoses that might interfere with the study (e.g. active peptic disease, inflammatory bowel disease), 5) a history of malignancy that might, to the best judgment of the doctor, interfere with the study, 6) any infectious or inflammatory disease within the last month, 7) active medically treated asthma, 8) baseline levels of HsCRP > 10mg/liter, 9) steroid treatment for any indication, 10) fecal incontinence, and 11) treatment with probiotics or antibiotics of any kind within the last 4 weeks, 11) Diabetes.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Symptom relief (abdominal pain and stool consistency) | 8 weeks
  Abdominal pain intensity, stool consistency, will be assessed by visual analogue scales (VAS) with scales from 0 (no symptom at all) to 10 (the worst possible symptom.
  The definition of treatment responders is based on the FDA Draft Guidance for Clinical Evaluation of Products for Treatment of Irritable Bowel Syndrome.
  * A Pain Intensity Responder is a patient who experiences a 30% or greater decrease in the weekly average of worst abdominal pain in past 24 hours in the past 24 hours compared to baseline.
  * A Stool Consistency Responder is a patient who has a greater than 50% decrease in the number of days with at least one stool ≥ type 6 using the Bristol Stool Scale (BSS).
  * A patient will be classified as an overall responder if they achieve the above improvement in pain intensity and stool consistency for at least 50 percent of the time.

SECONDARY OUTCOMES:
Improvement in other specific IBS symptoms, i.e., gas and bloating, feeling of urgency | 8 weeks
  Specific IBS symptoms, i.e., gas and bloating, feeling of urgency, will be assessed by visual analogue scales (VAS) with scales from 0 (no symptom at all) to 10 (the worst possible symptom).
Reduce hs-CRP levels | 8 weeks
  Blood will be drawn from IBS-D patients after a 12-hour fast and will be analyzed for hs-CRP.
Improve the cholinergic status | 8 weeks
  Plasma cholinesterase catalytic activity measurements will involve adaptation of a spectrophotometric method to a microtiter plate assay
Reduce calprotectin levels | 8 weeks
  At the beginning and at the end of the treatment period, fecal samples will be obtained for the measurement of calprotectin levels.
  The quantitative concentration of calprotectin will be determined by enzyme linked immunosorbent assay (ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: Ami Sperber, MD, Study Director — Tel Aviv Medical Center; Roy Dekel, MD, Principal Investigator — Tel Aviv Medical Center
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Central Israel, Israel